CLINICAL TRIAL: NCT05877625
Title: Study on Dynamic Environmental Exposome of ICU and the Establishment of Microbial Transmission Model Between Environment and Host
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Peking University Third Hospital (Other)
Collaborators: Zhejiang University (Other); Central South University (Other)
Responsible Party: Sponsor
Other Study IDs: M2022419
Record Dates: First submitted 2023-05-17; First posted 2023-05-26 (Actual); Last update posted 2023-06-22 (Actual); Status verified 2023-05

CONDITIONS: Hospital Acquired Infection; Ventilator-associated Pneumonia
Keywords: Environment exposure; Microbial Colonization; Microbiome
MeSH Terms: conditions — Cross Infection; Pneumonia, Ventilator-Associated; Communicable Diseases | interventions — Bronchoscopes

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 90 Days
Biospecimen Retention: Samples With DNA — endotracheal aspiration, bronchoalveolar lavage fluid
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (3):
- open ICU: open ICU: open ICU
  Interventions: Procedure: Expectoration care
- negative ICU: negative ICU: negative-pressure laminar flow ward
  Interventions: Procedure: Expectoration care
- positive ICU: positive ICU: laminar flow ward
  Interventions: Procedure: Expectoration care

INTERVENTIONS:
Procedure: Expectoration care — 1. Endotracheal aspiration: from discarded samples after expectoration care
  2. BALF (bronchoalveolar lavage fluid): if patients with fiber bronchoscope examination, take the rest of the BALF after examination
  3. Oropharyngeal swabs
  Other Names: Bronchoscope; Oropharyngeal swabs

SUMMARY:
HAI (Hospital-acquired infection) is very common in ICU，and lack of understanding of environmental exposure omics and environment-host microbial interactions restricts the prevention and control of HAI. In this project, the investigators try to analyze the spatial and temporal distribution characteristics and evolution of microorganisms and their functions in the ICU environment through metagenome.

DETAILED DESCRIPTION:
This observational study aims to analyze the spatial and temporal distribution characteristics and evolution of microorganisms and their functions in the ICU environment. The investigators will conduct weekly air microbiome sampling and microbiome sampling at 5 high-frequency contact points in different types of ICU units in three hospitals for one consecutive year, and collect dynamic pharyngeal swabs from ICU ward health care workers and dynamic clinical specimens (endotracheal aspiration, and bronchoalveolar lavage fluid) from patients with ventilator-associated pneumonia in ICU ward. With DNA high-throughput sequencing technology, the investigators will analyze the spatial and temporal distribution characteristics and evolution of microorganisms and their functions in the ICU environment, and provide support for HAI prevention.

ELIGIBILITY:
Inclusion Criteria:

* With mechanical ventilation
* Age ≥18 years
* Anticipated ICU stay for more than 2 days
* With two or more of the following ventilator-associated pneumonia (VAP) risk factors
* VAP risk factors: Age ≥ 60 years old; Patients with chronic lung disease; Long-term bedridden; Unconsciousness; Sputum is not easily coughed up; Antibiotics have been used before mechanical ventilation; Long-term use of H receptor blockers and proton pump inhibitors.

Exclusion Criteria:

* Patients who have not signed the informed consent
* Pregnant
* Systemic diseases and recent use of related drugs
* History of infectious diseases, such as tuberculosis or PPD positive
* History of hypertension and poor blood pressure control (SBP / DBP > = 140mmHg)
* With severe mental illness
* Long term use of traditional Chinese medicine, probiotics, gastric mucosal protective agents, proton pump inhibitors, chemotherapy or immunosuppressive drugs, etc.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with mechanical ventilation, age ≥18 years, anticipated ICU stay for more than 2 days, and with two or more of the following ventilator-associated pneumonia (VAP) risk factors were included in this study.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Actual)
Dates: Start 2022-08-01 (Actual); Primary Completion 2023-07-31 (Estimated); Study Completion 2023-08-31 (Estimated)

PRIMARY OUTCOMES:
Community of microbiome in ICU | 1 year
  the dynamic changes of metagenomic/16s sequencing data

CONTACTS AND LOCATIONS:
Locations (1):
- Peking University Third Hospital, Beijing, Beijing Municipality, China